CLINICAL TRIAL: NCT04932473
Title: ALFAsleep: Exploring Cognitive and Biological Correlates of Sleep Quality and Their Potential Links With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ALFAsleep-BBRC2018
Record Dates: First submitted 2021-06-08; First posted 2021-06-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cognitively Unimpaied

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main goal of this study is to perform a multimodal characterization of brain structural and functional changes, as well as changes in Alzheimer's disease (AD) biomarkers, as a function of sleep quality measures. Cross-sectional data will enable us to confirm and expand previous knowledge in a large and well-phenotyped population, while longitudinal data will allow us to test the hypothesis of the existence of a bidirectional relationship between sleep quality and AD.

DETAILED DESCRIPTION:
The main goal of this study is to perform a multimodal characterization of brain structural and functional changes, as well as changes in Alzheimer's disease (AD) biomarkers, as a function of sleep quality measures. Cross-sectional data will enable us to confirm and expand previous knowledge in a large and well-phenotyped population, while longitudinal data will allow us to test the hypothesis of the existence of a bidirectional relationship between sleep quality and AD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are currently participating in the ALFA+ study (cognitively healthy adults aged between 45-65 years at the moment of the inclusion in the 45-65/FPM2012 study).
* Subjects from whom CSF and/or neuroimaging biomarkers have been acquired during the last 36 months prior to their enrollment in the current study.

Exclusion Criteria:

* Presence of cognitive impairment.
* Presence of clinically relevant neurological disorder, psychiatric disorder or other medical conditions that may jeopardize the interpretation of the study results according to the investigator criteria
* For the PSG sub-study, participants currently treated with drugs that may interfere in PSG data interpretation (e.g. antidepressants or benzodiazepines).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 200 participants from the BBRC ALFA+ study (ALFA - FPM - 0311) will be selected based on their core AD biomarker profile to characterize their sleep quality with objective (actigraphy and RUSleeping RTS) and subjective measures.
  Participants will be classified into two different groups, based on previously established CSF biomarkers cut off values, as follows: 1) Controls: individuals with CSF Aβ42/ Aβ40 ratio > 0.071 ng/mL (considered as without altered AD biomarkers). 2) Preclinical AD: individuals with CSF Aβ42/ Aβ40 ratio 0.071 ≤ ng/mL (considered as with evidence of brain amyloidosis). However, it must be noted that thresholds for core biomarker abnormalities in preclinical AD, is an ongoing field of research and that these thresholds may vary with the addition of novel data/evidence resulting from our group and others.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Sleep quality | up to 2 weeks
  Actigraphy-derived sleep quality measures

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelonabeta Brain Research Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fauria K, Minguillon C, Knezevic I, Tort-Colet N, Stankeviciute L, Hernandez L, Radoi A, Deulofeu C, Fuentes-Julian S, Turull I, Fuste D, Sanchez-Benavides G, Arenaza-Urquijo EM, Suarez-Calvet M, Holst SC, Garces P, Mueggler T, Zetterberg H, Blennow K, Arqueros A, Iranzo A, Domingo Gispert J, Molinuevo JL, Grau-Rivera O. Exploring cognitive and biological correlates of sleep quality and their potential links with Alzheimer's disease (ALFASleep project): protocol for an observational study. BMJ Open. 2022 Dec 30;12(12):e067159. doi: 10.1136/bmjopen-2022-067159. PMID 36585141